CLINICAL TRIAL: NCT00475709
Title: An Observational, Prospective Evaluation of the Trifecta Valve
Brief Title: Aortic Valve Replacement With Trifecta(TM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0501
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Insufficiency; Regurgitation, Aortic Valve; Aortic Valve Incompetence; Aortic Valve Stenosis
Keywords: aortic valve; heart valve; tissue valve; bioprosthesis; valve disorder; valve disease; cardiac surgery; aortic valve stenosis; aortic valve regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trifecta Aortic Heart Valve (Experimental): All subjects enrolled into the study are implanted with the Trifecta Aortic Heart Valve.
  Interventions: Device: Trifecta Aortic Heart Valve

INTERVENTIONS:
Device: Trifecta Aortic Heart Valve — Surgical replacement of the aortic valve with the Trifecta Aortic Heart Valve.

SUMMARY:
To confirm the clinical safety and effectiveness of the Trifecta valve.

DETAILED DESCRIPTION:
The clinical investigation is a multi-center, multi-country, prospective, non-randomized, observational study designed to evaluate the safety and effectiveness of the Trifecta valve.

ELIGIBILITY:
Inclusion Criteria:

* Requires aortic valve replacement (heart surgery such as bypass is allowed at the same time).
* Legal age.
* Signed informed consent prior to surgery.
* Willing to complete all follow-up requirements.

Exclusion Criteria:

* Pregnant or nursing women.
* Have already had a valve replaced other than the aortic valve.
* Needs another valve replaced.
* Cannot return for required follow-up visits.
* Have active endocarditis.
* Acute preoperative neurological event (such as a stroke).
* Renal dialysis.
* History of substance abuse within one year, or a prison inmate.
* Participating in another study.
* Life expectancy less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartzell Schaff, MD, Principal Investigator — Mayo Clinic
Locations (18):
- United States (18):
  - USC Keck School of Medicine, Dept. of Cardiothoracic Surgery, USC University Hospital, Los Angeles, California
  - Sarasota Memorial Hospital/Clinical Research Center, Sarasota, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - NYU Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mission Hospitals, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Main Line Health Heart Center, Wynnewood, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Implanted With Trifecta Valve: All subjects enrolled into the study are implanted with the Trifecta Aortic Heart Valve.
Period: Overall Study
Arm/Group | Subjects Implanted With Trifecta Valve
Started | 1022
Eligible of Analysis | 1014 (Excludes eight ineligible subjects)
Completed | 946
Not Completed | 76
Not completed — Did not meet eligibility criteria | 8
Not completed — Death | 41
Not completed — Device Explant | 6
Not completed — Lost to Follow-up | 21

BASELINE CHARACTERISTICS:
Arm/Group | Trifecta Aortic Heart Valve
Number analyzed (Participants) | 1014
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364
  Male | 650

OUTCOME MEASURES:

1. Primary Outcome: Late Adverse Event Rates
Description: Late patient years are calculated from 31 days post-implant to the date of the last follow-up visits (or contact) or adverse events.
  Late Patient year calculation:[(Number of late adverse events/sum of late patient years) x 100]
Time Frame: Events occurring greater than or equal to 31 days post-implant.
Population: Analysis based on per protocol. Eight subjects did not meet eligibility criteria and were excluded from this analysis.
Measure: Number; unit: percentage of events/late patient years
Arm/Group | Trifecta Aortic Heart Valve
Number analyzed (Participants) | 1014
percentage of events/late patient years
  Thromboembolism | 1.90 [NA to NA]
  Valve Thrombosis | 0
  Major Bleed | 2.61
  Nonstructural Dysfunction | 0.12
  Endocarditis | 1.07
  Clinically Significant Hemolysis | 0.0
  Structural Deterioration | 0.12
  Valve Reoperation | 0.59
  Mortality (All Cause) | 2.72

2. Primary Outcome: Characterize Patient NYHA Functional Classification Status.
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest.
  The Criteria Committee of the New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th ed. Boston, Mass: Little, Brown & Co; 1994:253-256.
Time Frame: 1 year
Population: Analysis based on per protocol. Eight subjects did not meet eligibility criteria and were excluded from this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trifecta Aortic Heart Valve
Number analyzed (Participants) | 1014
percentage of participants
  NYHA I at 1 year | 85.3
  NYHA II at 1 year | 13.5
  NYHA III at 1 year | 1.2
  NYHA IV at 1 year | 0

3. Primary Outcome: Characterize the Hemodynamic Performance of the Valve.
Description: Gradient is the pressure difference from one side of the valve to the other side of the valve. For this study pressure is measured in mmHg.
  Mean gradient for each patient is the average of the pressure differences from one side of the valve to the other side of the valve.
  Mean gradient for each valve size (19mm, 21mm, 23mm, 25mm, 27mm, 29mm)is the average of the mean gradient for each patient with that valve size.
Time Frame: 1 year
Population: Analysis based on per protocol. Eight subjects did not meet eligibility criteria and were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Trifecta Aortic Heart Valve
Number analyzed (Participants) | 1014
mm Hg
  19 mm Mean Gradient (1 year) | 10.7 (4.6)
  21 mm Mean Gradient (1 year) | 8.1 (3.5)
  23 mm Mean Gradient (1 year) | 7.2 (2.8)
  25 mm Mean Gradient (1 year) | 6.2 (2.7)
  27 mm Mean Gradient (1 year) | 4.8 (2.0)
  29 mm Mean Gradient (1 year) | 4.7 (1.6)

ADVERSE EVENTS:
Description: Early (adverse events occuring on or before 30 days post procedure) and Late(adverse events occurring greater than or equal to 31 days post procedure) are combined for the Valve Related Serious Adverse Event data analysis.
Arm/Group | Subjects Implanted With Trifecta Valve
Serious Adverse Events (participants affected / at risk) | 147/1014
Other Adverse Events (participants affected / at risk) | 0/1014
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted With Trifecta Valve (N=1014)
Clinically Significant Hemolysis (Blood and lymphatic system disorders) | 0 (0)
Thromboembolism (Cardiac disorders) | 40 (43)
Valve Thrombosis (Cardiac disorders) | 0 (0)
Major Bleed (General disorders) | 96 (103)
Non-structural dysfunction (Cardiac disorders) | 4 (4)
Endocarditis (Infections and infestations) | 9 (9)
Structural deterioration (Cardiac disorders) | 1 (1)
Reoperation (Surgical and medical procedures) | 6 (6)
Valve related Mortality (Cardiac disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
The SAEs reported are based on the Edmunds criteria noted in Edmunds LH, Clark RE, Cohn LH, Grunkemeier GL, Miller CM, Weisel RD. Guidelines for reporting Morbidity and Mortality after Cardiac Valvular Operations. Ann Thorac Surg 1996;62:932-5.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other